CLINICAL TRIAL: NCT05814107
Title: A Double-Blind, Randomized, Placebo-Controlled Phase 1 Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Doses of CT-996 in Overweight/Obese Participants and in Patients With Type 2 Diabetes Mellitus
Brief Title: Phase 1 Study of CT-996 in Overweight/Obese Participants and Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Carmot Australia First Pty Ltd (Industry)
Collaborators: Carmot Therapeutics, Inc. (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Organization: Carmot Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CT-996-201
Record Dates: First submitted 2023-02-23; First posted 2023-04-14 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes; Overweight or Obesity
Keywords: Type 2 Diabetes; Obesity; Overweight
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Part 1: CT-996 SAD Cohort 1 (Experimental)
  Interventions: Drug: CT-996
- Part 1: CT-996 SAD Cohort 2 (Experimental)
  Interventions: Drug: CT-996
- Part 1: CT-996 SAD Cohort 3, Then SAD Cohort 5 (Experimental): During SAD Cohort 3, participants will be dosed under fasted conditions. During SAD Cohort 5, the same participants will receive the same dose under high-fat fed conditions.
  Interventions: Drug: CT-996
- Part 1: CT-996 SAD Cohort 4 (Experimental)
  Interventions: Drug: CT-996
- Part 1: CT-996 SAD Cohort 6 (Experimental)
  Interventions: Drug: CT-996
- Part 1: Placebo SAD Cohort (Placebo Comparator)
  Interventions: Drug: Placebo
- Part 2: CT-996 MAD Cohort 1 (Experimental)
  Interventions: Drug: CT-996
- Part 2: CT-996 MAD Cohort 2 (Experimental)
  Interventions: Drug: CT-996
- Part 2: CT-996 MAD Cohort 3 (Experimental)
  Interventions: Drug: CT-996
- Part 2: Placebo MAD Cohort (Placebo Comparator)
  Interventions: Drug: Placebo
- Part 3: CT-996 MD T2DM Cohort 1 (Experimental)
  Interventions: Drug: CT-996
- Part 3: CT-996 MD T2DM Cohort 2 (Experimental)
  Interventions: Drug: CT-996
- Part 3: Placebo MD T2DM Cohort (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CT-996 — Capsule of CT-996
  Other Names: RO7795081; RG6652
  Arms: Part 1: CT-996 SAD Cohort 1; Part 1: CT-996 SAD Cohort 2; Part 1: CT-996 SAD Cohort 3, Then SAD Cohort 5; Part 1: CT-996 SAD Cohort 4; Part 1: CT-996 SAD Cohort 6; Part 2: CT-996 MAD Cohort 1; Part 2: CT-996 MAD Cohort 2; Part 2: CT-996 MAD Cohort 3; Part 3: CT-996 MD T2DM Cohort 1; Part 3: CT-996 MD T2DM Cohort 2
Drug: Placebo — Capsule of placebo matching CT-996.
  Arms: Part 1: Placebo SAD Cohort; Part 2: Placebo MAD Cohort; Part 3: Placebo MD T2DM Cohort

SUMMARY:
This study is designed to assess the safety and tolerability, pharmacokinetics, and pharmacodynamics of CT-996 in overweight/obese participants and participants with Type 2 Diabetes Mellitus (T2DM).

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled, dose escalation, first in human study designed to assess the safety and tolerability, pharmacokinetics, and pharmacodynamics of CT-996 when administered as single ascending doses (SAD) and multiple-ascending doses (MAD) in overweight/obese participants and as multiple doses (MD) in patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Participants 18-65 years old, inclusive
* BMI of 25 - 40, inclusive
* Stable body weight for two months

Additional Inclusion Criterion for Part 3 (MD T2DM cohorts) only:

* Participants in Part 3 should have a documented diagnosis of Type 2 Diabetes Mellitus (T2DM)
* Participants in Part 3 should have glycated hemoglobin (HbA1c) between 7.0% and 10.0%

Exclusion Criteria:

* History of significant medical conditions and malignancy
* Uncontrollable hypertension
* History of alcoholism or drug addiction within 1 year prior to Screening
* Current or recent participation in an investigational clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From first study drug administration until last safety follow-up (up to 31 days [Part 1] or 58 days [Parts 2 and 3])

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of CT-996 | At prespecified timepoints from Day 1 to Day 5 (Part 1) or Day 33 (Parts 2 and 3)
Time to Maximum Observed Plasma Concentration (Tmax) of CT-996 | At prespecified timepoints from Day 1 to Day 5 (Part 1) or Day 33 (Parts 2 and 3)
Area Under the Concentration-Time Curve (AUC) from Time 0 to the Time of Last Measurable Concentration (AUC0-t) of CT-996 | At prespecified timepoints from Day 1 to Day 5 (Part 1) or Day 33 (Parts 2 and 3)
AUC from Time 0 Extrapolated to Infinity (AUC0-inf) of CT-996 | At prespecified timepoints from Day 1 to Day 5 (Part 1) or Day 33 (Parts 2 and 3)
Apparent Terminal Elimination Half-Life (t1/2) of CT-996 | At prespecified timepoints from Day 1 to Day 5 (Part 1) or Day 33 (Parts 2 and 3)
Part 1 Cohorts: Clearance (CL) of CT-996 | At prespecified timepoints from Day 1 to Day 5
Part 1 Cohorts: Volume of Distribution (V) of CT-996 | At prespecified timepoints from Day 1 to Day 5
Part 2 Cohorts: Minimum Observed Plasma Concentration (Cmin) of CT-996 | At prespecified timepoints from Day 1 to Day 33
Parts 2 and 3 Cohorts: Clearance Divided by the Bioavailable Fraction (CL/F) of CT-996 | At prespecified timepoints from Day 1 to Day 33
Parts 2 and 3 Cohorts: Volume of Distribution Divided by the Bioavailable Fraction (Vz/F) of CT-996 | At prespecified timepoints from Day 1 to Day 33
Part 1 SAD Cohorts 3 and 5: Food Effect of a High-Fat Meal on Cmax of CT-996 | At prespecified timepoints for up to 14 days
  Determine the effect of a high-fat meal on the PK of CT-996 following a single dose
Part 1 SAD Cohorts 3 and 5: Food Effect of a High-Fat Meal on AUC of CT-996 | At prespecified timepoints for up to 14 days
  Determine the effect of a high-fat meal on the PK of CT-996 following a single dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Carmot Therapeutics, Inc., a Member of the Roche Group
Locations (2):
- Nucleus Network Pty Ltd., Melbourne, Australia
- Avant Santé Research Center S.A. de C.V., San Pedro Garza García, Mexico

IPD SHARING:
Plan to Share IPD: No